CLINICAL TRIAL: NCT05661786
Title: Clinical Outcomes of HBeAg-negative Chronic Hepatitis B Patients With Indeterminate Phase: a Multi-center, Prospective, Observational Cohort Study (PILOT)
Brief Title: Clinical Outcomes of HBeAg-negative CHB Patients With Indeterminate Phase
Acronym: PILOT
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Chao Wu, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: NJDTID-2201
Record Dates: First submitted 2022-08-13; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic hepatitis b; Indeterminate phase; hepatitis B surface antigen clearance; Hepatocellular carcinoma; Antiviral treatment
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation cohort
  Interventions: Other: Observation
- Treatment cohort
  Interventions: Other: Antiviral treatment

INTERVENTIONS:
Other: Observation — Monitor every 6 months
  Groups: Observation cohort
Other: Antiviral treatment — Receive first-line antiviral treatment, including entecavir, tenofovir disoproxil fumarate, tenofovir alafenamide, tenofovir amibufenamide or peginterferon
  Groups: Treatment cohort

SUMMARY:
Chronic hepatitis B virus (HBV) infection remains a global public health burden around the world. Investigating the disease process of chronic hepatitis B (CHB) is essential to individual management in clinical practice. According to American Association for the Study of Liver Diseases (AASLD) 2018 Hepatitis B Guidance, CHB can be classified into four phases: immune-tolerant CHB, HBeAg-positive immune active CHB, inactive CHB and hepatitis B e antigen (HBeAg)-negative immune active CHB. Antiviral therapy is recommended in patients with HBeAg-positive or -negative immune active CHB patients to reduce the incidence of liver cirrhosis and hepatocellular carcinoma, while periodic monitoring is recommended for inactive carrier and immune-tolerant CHB patients. However, a substantial proportion of patients fall into an indeterminate phase whose serum HBV DNA and alanine aminotransferase levels do not fit well into these well-described phases. Most of CHB patients with indeterminate phase are HBeAg negative. However, the clinical outcomes of these patients remain unclear. Therefore, the purpose of this study is to investigate the clinical outcomes of HBeAg-negative chronic hepatitis B patients with indeterminate phase.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatitis B surface antigen (HBsAg) positive over 6 months
2. Age ≥18 years
3. Treatment-naïve
4. HBeAg negative, anti-HBe positive
5. HBV DNA >2000 IU/mL
6. Persistently normal alanine transaminase (ALT)
7. Liver inflammation <G2 or A2 and liver fibrosis <S2 or F2 before enrollment, or liver stiffness >8 kilopascals (kPa)
8. No family history of liver cirrhosis or hepatocellular carcinoma

Exclusion Criteria:

1. Coinfection with hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus or human immunodeficiency virus;
2. Coexisting of hepatocellular carcinoma and other malignancy, or alpha-fetoprotein >upper limit of normal at enrollment;
3. Presence of liver cirrhosis;
4. Alcohol abuse within the last year (ethanol: male >40 g/d, female >20 g/d; or heavy drinking within 2 weeks before enrollment: ethanol >80 g/d), or history of drug abuse;
5. Participating in other clinical trials in the last 3 months;
6. Coexisting of autoimmune liver diseases;
7. Pregnant or planned pregnancy in a short term or lactation patients;
8. History of severe heart disease, mental disease;
9. Uncontrolled diabetes, hypertension, thyroid dysfunction, retinopathy, autoimmune diseases;
10. Neutrophil count <2×10^9/L and/or platelet count <100×10^9/L;
11. History of organ transplantation or preparing for organ transplantation;
12. Using immunosuppressive drugs;
13. Undergone organ transplantation or preparing for organ transplantation;
14. Receiving immunosuppressive agents;
15. Patients thought by the investigators not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-negative chronic hepatitis B patients with indeterminate phase
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of hepatocellular carcinoma at 240 weeks | 240 weeks
The HBsAg clearance rate at 240 weeks | 240 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Third Hospital of Changzhou, Changzhou, Jiangsu
  - Huai'an No.4 People's Hospital, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Suqian People's Hospital, Suqian, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu J, Liang W, Jing W, Liu M. Countdown to 2030: eliminating hepatitis B disease, China. Bull World Health Organ. 2019 Mar 1;97(3):230-238. doi: 10.2471/BLT.18.219469. Epub 2019 Jan 28. PMID 30992636
- [Result] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Result] Huang DQ, Li X, Le MH, Le AK, Yeo YH, Trinh HN, Zhang J, Li J, Wong C, Wong C, Cheung RC, Yang HI, Nguyen MH. Natural History and Hepatocellular Carcinoma Risk in Untreated Chronic Hepatitis B Patients With Indeterminate Phase. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1803-1812.e5. doi: 10.1016/j.cgh.2021.01.019. Epub 2021 Jan 16. PMID 33465482
- [Result] Yao K, Liu J, Wang J, Yan X, Xia J, Yang Y, Wu W, Liu Y, Chen Y, Zhang Z, Li J, Huang R, Wu C. Distribution and clinical characteristics of patients with chronic hepatitis B virus infection in the grey zone. J Viral Hepat. 2021 Jul;28(7):1025-1033. doi: 10.1111/jvh.13511. Epub 2021 Apr 26. PMID 33797145
- [Result] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Result] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Result] Bonacci M, Lens S, Marino Z, Londono MC, Rodriguez-Tajes S, Mas A, Garcia-Lopez M, Perez-Del-Pulgar S, Sanchez-Tapias JM, Forns X. Anti-viral therapy can be delayed or avoided in a significant proportion of HBeAg-negative Caucasian patients in the Grey Zone. Aliment Pharmacol Ther. 2018 May;47(10):1397-1408. doi: 10.1111/apt.14613. Epub 2018 Mar 25. PMID 29577350
- [Result] Choi GH, Kim GA, Choi J, Han S, Lim YS. High risk of clinical events in untreated HBeAg-negative chronic hepatitis B patients with high viral load and no significant ALT elevation. Aliment Pharmacol Ther. 2019 Jul;50(2):215-226. doi: 10.1111/apt.15311. Epub 2019 May 28. PMID 31135074